CLINICAL TRIAL: NCT03306641
Title: A One-Week Crossover Dispensing Evaluation of Gemini Daily Wear Soft Contact Lenses
Brief Title: A One-Week Crossover Dispensing Evaluation of New Daily Wear Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CV-17-29
Record Dates: First submitted 2017-08-15; First posted 2017-10-11 (Actual); Results first posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: This will be a double-masked, bilateral, 1-week crossover, dispensing study, comparing the test daily wear lens against nelfilcon A control lens, such that each lens type will be worn for 1 week each. Each subject will be randomized to wear either the test lenses or the control lenses as a matched pair.
Who Masked: Participant, Investigator
Masking Description: The contact lenses coding will be masked to both the investigator and subject. If standard labeling does not sufficiently mask the study material then over-labeling will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Test Contact Lens (Active Comparator): Per randomized schedule, subject will wear a pair of the test lens or control lens for one week and then cross-over with the control pair for 1 week.
  Interventions: Device: Test Contact Lens; Device: Nelfilcon A
- nelfilcon A lens (control) (Active Comparator): Per randomized schedule, subject will wear a pair of the control lens for one week and then cross-over with the test pair for 1 week.
  Interventions: Device: Test Contact Lens; Device: Nelfilcon A

INTERVENTIONS:
Device: Test Contact Lens — Daily disposable contact lens
Device: Nelfilcon A — Focus Dailies All Day Comfort contact lens (nelfilcon A)

SUMMARY:
The purpose of this study is to validate the clinical performance of a new contact lens design when worn over a period 1 week compared to nelfilcon A (control).

DETAILED DESCRIPTION:
The purpose of this study is to validate the clinical performance of a new contact lens design when worn over a period of 1 week compared to nelfilcon A (control). The primary outcomes of interest is lens fit acceptance.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age and has full legal capacity to volunteer.
* Is no greater than 55 years of age.
* Has read and understood the information consent letter.
* Is willing and able to follow instructions and maintain the appointment schedule.
* Is an adapted soft contact lens wearer having worn lenses for a minimum of 4 weeks prior to the study.
* Has spectacle cylinder ≤1.00D in both eyes.
* Has spherical contact lens power requirement between -1.00D and -6.00D in both eyes.
* Has manifest refraction visual acuities (VA) equal to or better than logMAR equivalent of 20/25 in each eye.
* Wears CLs in both eyes (monvision acceptable, but not monofit)
* Has clear corneas and no active ocular disease.
* Has not worn lenses for at least 12 hours before the examination.
* Is willing to wear the study contact lenses for a minimum 8 hours per day/6 days per week

Exclusion Criteria:

* Has never worn contact lenses before.
* Has any systemic disease affecting ocular health.
* Is using any systemic or topical medications that will affect ocular health.
* Has any ocular pathology or severe insufficiency of lacrimal secretion (moderate to severe dry eyes) that would affect the wearing of contact lenses.
* Has persistent, clinically significant corneal or conjunctival staining using sodium fluorescein dye.
* Has any clinically significant lid or conjunctival abnormalities, active neovascularization or any central corneal scars.
* Is aphakic.
* Has strabismus/amblyopia.
* Has undergone corneal refractive surgery.
* Is pregnant, lactating or planning a pregnancy.
* Is participating in any concurrent clinical or research study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Optics Research Lab (CORL) Indiana University School of Optometry, Indiana University, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Contact Lens Then Nelfilcon A Lens (Control): Per randomized schedule, subject will wear a pair of the test lens for one week and then cross-over with the control pair for 1 week.
  Test Contact Lens: Daily disposable contact lens
  Nelfilcon A: Focus Dailies All Day Comfort contact lens (nelfilcon A)
- Nelfilcon A Lens (Control) Then Test Contact Lens: Per randomized schedule, subject will wear a pair of the control lens for one week and then cross-over with the test pair for 1 week.
  Test Contact Lens: Daily disposable contact lens
  Nelfilcon A: Focus Dailies All Day Comfort contact lens (nelfilcon A)
Period: First Intervention
Arm/Group | Test Contact Lens Then Nelfilcon A Lens (Control) | Nelfilcon A Lens (Control) Then Test Contact Lens
Started | 23 | 22
Completed | 23 | 22
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Test Contact Lens Then Nelfilcon A Lens (Control) | Nelfilcon A Lens (Control) Then Test Contact Lens
Started | 23 | 22
Completed | 23 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Per randomized schedule, subject will wear either a pair of the test lens or control lens for one week and then cross-over to the other pair for 1 week.
  Test Contact Lens: Daily disposable contact lens
  Nelfilcon A: Focus Dailies All Day Comfort contact lens (nelfilcon A)
Arm/Group | Overall Study
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Lens Fit Acceptance
Description: Overall lens fit acceptance was measured on a scale of 0-4 in 0.25 steps (0=can't be worn, 1=Poor, 2=Fair, 3=Good, 4=Optimum)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Test Contact Lens: Per randomized schedule, subject will wear a pair of the test lens for one week in this cross-over study.
  Test Contact Lens: Daily disposable contact lens
- Nelfilcon A Lens (Control): Per randomized schedule, subject will wear a pair of the control lens for one week in this cross-over study.
  Nelfilcon A: Focus Dailies All Day Comfort contact lens (nelfilcon A)
Arm/Group | Test Contact Lens | Nelfilcon A Lens (Control)
Number analyzed (Participants) | 45 | 45
units on a scale | 2.6 (0.6) | 3.1 (0.3)

2. Primary Outcome: Lens Fit Acceptance
Description: as for outcome 1
Time Frame: 1-Week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Contact Lens | Nelfilcon A Lens (Control)
Number analyzed (Participants) | 45 | 45
units on a scale | 2.6 (0.6) | 3.0 (0.4)

ADVERSE EVENTS:
Time Frame: From dispense up to 1-week on each pair of lenses, a total of two weeks.
Arm/Group | Test Contact Lens | Nelfilcon A Lens (Control)
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT03306641/Prot_SAP_000.pdf